CLINICAL TRIAL: NCT00386880
Title: Prevalence of Phonophobia and Cutaneous Allodynia in Episodic Migraineurs
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: AA-Phono-CA
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Sound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with episodic migraine with allodynia: These are subjects with episodic migraine with allodynia
  Interventions: Other: Sounds
- Subjects with episodic migraine without allodynia: Subjects with episodic migraine without allodynia
  Interventions: Other: Sounds

INTERVENTIONS:
Other: Sounds

SUMMARY:
Cutaneous allodynia is an increased skin sensitivity experienced during a headache. It has been noted in several studies that in patients with migraine, seventy nine percent of the patients experienced allodynia on the facial skin on the same side as the headache. Understanding more about the occurrence of phonophobia (increased sensitivity to sound) and allodynia may help us understand how the pain system works in migraine. It is hoped that the knowledge gained from this trial may enable us to more effectively treat patients with migraine headache.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for migraine subjects:

* Age: 18 - 65 years, inclusive.
* Gender: male or female
* Diagnosis: Episodic migraine with or without aura, as defined by the International Headache Society (IHS), for at least 6 months prior to enrollment.
* An average of ≥1 migraine attack per month over the 6-month period prior to enrollment.
* An average of <15 headache (of any type) days per month for the 6 months prior to enrollment.
* Normal audiogram. (A hearing threshold of 20 dB or less at the frequency range of 200-8000Hz.).

Inclusion criteria for control subjects:

* Age: 18 - 65 years, inclusive.
* Gender: male or female
* Non-headache sufferers with the exception of infrequent ETTH according to IHS criteria (lifetime occurrence of at least 10 episodes occurring on <1 day per month on average and <12 days per year)
* Normal audiogram, (A hearing threshold of 20 dB or less at the frequency range of 200-8000Hz.).

Exclusion criteria for migraine subjects:

* Any other headache diagnosis (e.g. cluster headache, hemicrania continua, post traumatic headache, etc.) except for episodic tension type headache (ETTH) with an average of no more than 10 ETTH headache days per month for the 6 months prior to enrollment (note: average <15 total HA days is specified in inclusion)
* Use of any headache preventive drug (determined by investigator) in the 90 days prior to screening.
* Treatment with botulinum toxin (for any indication) within the 90 day period prior to enrollment.
* Treatment with occipital nerve block or block, or block of any other nerve in the head or neck area, within the 30 day period prior to enrollment.
* Any dermatological disease that may affect skin sensation.
* Any neurological disease that may affect sensory functions (e.g stroke, multiple sclerosis, peripheral neuropathy).
* Cognitive disturbance that may affect the subject's ability to understand the study procedure.
* Significant psychiatric disturbance that may impair the subject from co-operating with the study procedures.
* Use of acute pain medications on a daily or frequent pattern (for any indication) as defined by the IHS.

Exclusion criteria for control subjects:

* Any other headache diagnosis except for IHS-defined infrequent ETTH.
* Use of any headache preventive drug (determined by investigator) in the 90 days prior to screening.
* Treatment with botulinum toxin (for any indication) within the 90 day period prior to enrollment.
* Treatment with occipital nerve block or block, or block of any other nerve in the head or neck area, within the 30 day period prior to enrollment.
* Any dermatological disease that may affect skin sensation.
* Any neurological disease that may affect sensory functions (e.g stroke, multiple sclerosis, peripheral neuropathy).
* Cognitive disturbance that may affect the subject's ability to understand the study procedure.
* Significant psychiatric disturbance that may impair the subject from co-operating with the study procedures.
* Use of acute pain medications on a daily or frequent pattern (for any indication) as defined by the IHS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women and men with a diagnosis of episodic migraine
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham A. Ashkenazi, M.D., Principal Investigator — Thomas Jefferson University
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Ashkenazi A, Yang I, Mushtaq A, Oshinsky ML. Is phonophobia associated with cutaneous allodynia in migraine? J Neurol Neurosurg Psychiatry. 2010 Nov;81(11):1256-60. doi: 10.1136/jnnp.2009.198481. Epub 2010 Jun 20. PMID 20562466

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Episodic Migraine With Allodynia: These are the subjects with episodic migraine with allodynia.
- Subjects With Episodic Migraine Without Allodynia: These are the subjects with episodic migraine without allodynia.
Period: Overall Study
Arm/Group | Subjects With Episodic Migraine With Allodynia | Subjects With Episodic Migraine Without Allodynia
Started | 30 | 8
Completed | 30 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects With Episodic Migraine: Subjects with less than 8 distict migraine episodes per month.
Arm/Group | Subjects With Episodic Migraine
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Phonophobia (Sound Sensitivity) and Allodynia (Skin Sensitivity) in Subjects With Episodic Migraine
Description: Measurement of phonophobia: determine sound aversion threshold (SAT), measured in dB during a migraine attack in subjects with and in subjects without allodynia.
Time Frame: Subjects with or without allodynia return during a migraine attack and are tested for Phonophobia.
Measure: Number; unit: participants
Groups:
- Subjects With Episodic Migraine Without Allodynia: These are subjects with episodic migraine without allodynia
Arm/Group | Subjects With Episodic Migraine With Allodynia | Subjects With Episodic Migraine Without Allodynia
Number analyzed (Participants) | 30 | 8
participants | 27 | 6
Statistical Analysis 1: Comparison: Subjects With Episodic Migraine With Allodynia vs Subjects With Episodic Migraine Without Allodynia; During the acute migraine attack, 90% of allodynic subjects and 75% of subjects without allodynia had phonophobia; Test type: Superiority or Other; p = 0.59, Fisher Exact — Fisher's exact test

ADVERSE EVENTS:
Arm/Group | Subjects With Episodic Migraine
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes